CLINICAL TRIAL: NCT01575886
Title: Enhancing Teachable Moment Communication for Smoking Cessation and Weight
Brief Title: Enhancing Teachable Moment Communication for Smoking Cessation and Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Susan Flocke, Associate Professor of Family Medicine and Community Health, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01CA105292_ETM; R01CA105292 (NIH)
Record Dates: First submitted 2012-04-06; First posted 2012-04-12 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Clinician Patient Communication; Smoking Cessation; Weight Management
Keywords: clinician patient communication; smoking cessation; weight management; primary care; health behavior change advice
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking cessation intervention (Experimental): This group receives the teachable moment communication process intervention focused on smoking cessation and contributes data at baseline (Time 1) and post intervention (Time 2).
  Interventions: Other: Teachable Moment Communication Process
- Delayed intervention group (Other): This group serves as the comparison group for the evaluation of the smoking cessation intervention at Time 1 and Time 2 data collection to complete the group randomized trial. This group of clinicians then has Time 3 data collection focused on weight management receives a revised intervention focused on teachable moment communication for weight management and has Time 4 data collected to evaluate the teachable moment for weight management training as a pre-post design.
  Interventions: Other: Teachable Moment Communication Process

INTERVENTIONS:
Other: Teachable Moment Communication Process — The Teachable Moment Communication Process intervention is designed to teach clinicians: (1) the skills necessary to recognize and foster teachable moments in clinical encounters, (2) strategies to effectively elicit the patients' perspective on health behavior change, and express their alignment with that perspective, and (3) the ability to respond to the patient in a non-confrontational manner while providing brief advice appropriate to the patient's expressed level of readiness to change. The Teachable Moment Communication Process intervention consists of two, 3-hour educational training sessions including didactic presentation, skill demonstration through video examples, skills practices with standardized patients, and feedback from peers and the trainers.

SUMMARY:
The goal of this study is to test an intervention that teaches clinicians to integrate the use of 'teachable moments' with the key skills of motivational interviewing tailored to address smoking and weight management in the primary care outpatient visit setting.

DETAILED DESCRIPTION:
A large burden of cancer morbidity and mortality is potentially preventable by changes in personal health behaviors. Health behavior advice (HBA) by primary care physicians, who provide basic health care to most Americans, holds great promise as a strategy to alter cancer-related health behaviors and to reduce morbidity and mortality. One potentially powerful strategy is the use of illness visits as a 'teachable moment'(TM) for health behavior change. Our in-depth analysis of audio recorded physician-patient interactions has led to new discoveries of the communication elements of a TM. First, effective TM's involve linking a health behavior to a salient patient problem and positioning the health behavior as a problem. Persuasion is accomplished by suggesting that changing the health behavior will improve the patient's salient concern. If done skillfully, the patient accepts the portrayal of the health behavior as a relevant problem and exhibits uptake of the health behavior change talk, possibly expressing a commitment to change. Our data reveal that TMs occur in 20% of health behavior discussions between physician and patient. More frequent (43%) , however, are TM 'attempts' which fail to engage the patient. These attempts lack two essential aspects of good patient-centered advice 1) eliciting the patient's readiness to change and 2) responding in alignment with the patient's expressed stage of change. We also observed 'missed opportunities' (20%) where the health behavior advice failed to link to a salient patient concern.

Therefore, the goal of this randomized trial is to test an intervention that teaches clinicians to integrate the use of TMs with the key skills of motivational interviewing tailored to address smoking and weight management in the outpatient visit setting. This goal will be accomplished using a group randomized trial of 32 clinicians (1152 patients). The initial Teachable Moment Communication Process (TMCP) intervention will focus on smoking cessation as the health behavior topic. After the initial intervention is evaluated, the clinicians assigned to the control group will receive a revised TMCP intervention with a focus on weight management. The TMCP intervention involves multiple modalities including skills-based training, practice with standardized patients and on-site coaching. Audio recordings of visits with patients who smoke or are obese will be used to assess both intervention and control clinicians' health behavior change strategies at baseline and post intervention. Patient surveys will be used to assess the effect of the observed health behavior change strategies on immediate and short-term patient outcomes. Leveraging clinicians' naturally-occurring health behavior change strategies by fostering the development of more effective communication skills has great potential to enhance patient health behavior change. This study will test this strategy and generate rich data about its effectiveness and how it is tailored by physicians in practice for both smoking and weight management; two important risk factors for cancer and other devastating chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting a clinician participating in the study on data collection days.
* For data collection Time 1 and 2, patients who report smoking at least 1 cigarette per day.
* For data collect times 3 and 4, patients who have a BMI > 30 or patients who have a BMI >25 and self-reporting any one of the following chronic conditions: high blood pressure, high cholesterol, heart disease or diabetes.

Exclusion Criteria:

* Inability to comprehend the invitation to participate in the study in English or Spanish
* No access to a telephone and no mailing address to complete follow up surveys.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
performance of the elements of the teachable moment communication process | evaluated at time of observed/audio recorded visit; visits are evaluated between 2 weeks and 3 months after clinician exposure to the educational intervention
  Analysis of the audio recorded visit is used to assess the performance of each of the key elements of the teachable moment communication process.
incremental behavior change for smoking | 6 weeks
  A 15-item self report measure of small behavior changes antecedent to smoking cessation. The measure is assessed prior to the visit and then 6-weeks after the observed visit and a change score is computed.

SECONDARY OUTCOMES:
duration of the visit | immediate
  the amount of time spent face to face with the clinician during the observed visit.

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Flocke, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Flocke SA, Antognoli E, Step MM, Marsh S, Parran T, Mason MJ. A Teachable Moment Communication Process for smoking cessation talk: description of a group randomized clinician-focused intervention. BMC Health Serv Res. 2012 May 3;12:109. doi: 10.1186/1472-6963-12-109. PMID 22554310